CLINICAL TRIAL: NCT03747822
Title: Evaluation of Soft Tissue Profile Changes Following Autogenous Fat or Onlay Polyetheretherketone(PEEK) Augmentation Versus Sliding Genioplasty for Correction of Deficient Chin
Brief Title: Evaluation of Soft Tissue Profile Changes Following Autogenous Fat or Onlay Polyetheretherketone (PEEK) Augmentation Versus Sliding Genioplasty for Correction of Deficient Chin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, asmaa mohmed helmy, assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20687
Record Dates: First submitted 2018-11-17; First posted 2018-11-20 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Patients With Deficient Chin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: a third party oral surgery specialist will be asked to assess the study participate according to a standardized assessment tool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- autogenous fat (Active Comparator): autogenous fat augmentation in deficient chin will be harvested from lower abdomen,inner or outer thigh
  Interventions: Procedure: fat filler,PEEK,sliding genioplasty
- PEEK (Active Comparator): Will use onlay PEEK augmentation in deficient chin.Virtual planning will be done using mimics software. A virtual osteotomy of the chin will be performed at the inferior border of the mandible same alignments as sliding genioplasty, then segmentation of the chin area will be done and according to the soft tissue analysis adjustment will be performed.
  Interventions: Procedure: fat filler,PEEK,sliding genioplasty
- Osseous sliding genioplasty (Other): Under general anesthesia, the preparation and the incision line will be performed same as PEEK augmentation .After complete exposure of the bone repositioning of the chin will be performed. Finally fixation will be obtained using x shape titanium plate.
  Interventions: Procedure: fat filler,PEEK,sliding genioplasty

INTERVENTIONS:
Procedure: fat filler,PEEK,sliding genioplasty — The procedure will be done under general anesthesia; the donor site lower abdomen, flank, lateral thigh, or inner thigh will be infused using a solution that consisted of 100 ml of normal saline with 50 mg (0.05%) of lidocaine and 0.1 ml of epinephrine. Liposuction will be performed using a 2-mm blunt cannula. A 20-cc syringe will be used to collect the fat. The fat will be injected into the chin in a supraperiosteal (subcutaneous) plane with a blunt 2-mm cannula using a fanning technique.

SUMMARY:
Fat is a filler with ideal properties as it naturally integrates into tissues with 100 % biocompatibility. Moreover, fat contains different cell types, including adipocytes, fibroblasts, smooth muscle cells, endothelial cells, and adipogenic progenitor cells called"preadipocytes"2, adipose-derived stem cells (ASCs) which have a differentiation potential similar to that of other mesenchymal stem cells and it could be harvested in great amounts with minimal donor-site morbidity, ASCs have proved to be particularly promising for regenerative therapies. In addition, it's relatively inexpensive and readily available, which makes it an attractive alternative for facial augmentation.

On the other hand PEEK is considered a highly biocompatible material with mechanical properties almost similar to cortical bone. It is widely used in cranioplasties and facial reconstruction.

DETAILED DESCRIPTION:
The chin is the most noticeable facial structure which plays an important role in perception of facial esthetics; therefore deficient chin is considered an annoying defect for the patient. Traditional techniques used for correction, which are osseous genioplasty and alloplastic augmentation, have some reported complications. These complications include hematoma in the floor of the mouth; though a rare complication is considered to be a life threatening condition. Also, wound dehiscence, infection, Chin hypoesthesia/dysesthesia due to mental nerve injury which occurs in 3.4% to 12% of cases , chin ptosis, lip ptosis, drooling, and an increase in lower teeth show due to failure to reattach the mentalis muscle to its natural origin on the anterior face of the mandibular body and tooth root damage which may occur during the osteotomy. Also bone resorption, implant displacement, infection and foreign body reaction were reported as a complication with some alloplastic implants .

This study aims to avoid the complications of surgical correction of deficient chin by using less invasive approach.

Trial design:

3 Groups of patients will be assigned to this trial: Study group1: Will use autogenous fat augmentation in deficient chin. Study group2: Will use onlay PEEK augmentation in deficient chin. Control group: Surgical correction of deficient chin with sliding genioplasty. Trial design: Randomized Controlled clinical Trial

ELIGIBILITY:
Inclusion Criteria:

•.Medically free patients.

* Patients with deficient chin..
* Age range is between 18 and 45 years
* No sex predilection.

Exclusion Criteria:

* Patients with systemic condition contraindicating with the surgical procedure.
* Previously corrected chin.
* Patients indicated for other skeletal mandibular procedure during the same surgical session.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
soft tissue analysis | year follow up
  assessment of soft tissue profile changes using computerized software ,land marks will be determined on soft tissue mask of patient's cone beam computed tomography (cbct) .The Frankfort horizontal (FH) plane will be chosen as a reference line .Horizontal soft tissue changes will be recorded parallel to the FH line and perpendicular on the nasion vertical (NV), whereas the vertical soft tissue changes will be recorded parallel to the NV and perpendicular on the FH line.The advancement will be measured by the change in the position of point Pg preoperatively and postoperatively (T2) from the NV line.The points (Pg, Pg', Me, Me', and B) will be measured for vertical and horizontal movements by a line from each point and perpendicular to the NV and the FH

IPD SHARING:
Plan to Share IPD: Undecided